CLINICAL TRIAL: NCT03643263
Title: Exploring the Relationship Between pH of Exhaled Breath Condensate and Disease Severity as Well as Prognosis of Bronchiectasis
Brief Title: Exhaled Breath Condensate Assessment in Stable Non-Cystic Fibrotic Bronchiectasis
Status: Completed | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Director, Head of respiratory medicine, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 20180323
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collected exhaled breath condensate specimens for pH test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The measurement of markers in the expired breath condensate has proven to be a useful method for assessing and monitoring airway inflammation. The aim of this study is to determine the amounts of pH in the expired breath condensate of patients with bronchiectasis, and the relationship between pH and the severity of bronchiectasis.

DETAILED DESCRIPTION:
The aim of this study is to determine the amounts of pH in the expired breath condensate of patients with bronchiectasis, and the relationship between pH and the severity of bronchiectasis. Further clarify the link between EBC pH and the risk of future acute exacerbations, mortality and lung function decline through a one-year follow-up. Hoping to explore new validated biomarkers of the disease severity and progression in bronchiectasis. During the observation, EBC pH and other valid indicators will be measured when patients were enrolled.

ELIGIBILITY:
Inclusion Criteria:Each subject must meet all of the following criteria to be included in this study:

1. Willing to join in and sign the informed consent form.
2. Age>18 years, the diagnosis of bronchiectasis need reference to the definition of "non-cystic fibrosis bronchiectasis guideline" published by British Thoracic Society in 2010 or 2012 China bronchiectasis expert consensus, clinical symptoms of cough and expectoration, with or without intermittent hemoptysis, and chest CT showed bronchiectasis there.
3. All patients were clinically stable and had no evidence of infection or acute infective exacerbation (lower or upper respiratory tract) for at least 4 weeks before the study.
4. Patients with good compliance: the subject must be willing to follow the test plan requirements in the research center to complete all the assessment of the visit.

Control Subjects:

1. All normal subjects had a negative history of allergy (negative skin prick tests to common allergens);
2. Normal lung function, and normal bronchial reactivity.
3. No history of any lung disease (except for the history of pneumonia in the past time and small pulmonary nodules).

Exclusion Criteria:Subjects who meet any of the following criteria should be excluded from this study:

1. Patients with a history of other respiratory diseases (cystic fibrosis, allergic bronchopulmonary aspergillosis, asthma, 1-antitrypsin deficiency, pulmonary tuberculosis, COPD, lung cancer, interstitial lung disease)and atopic diseases were excluded；
2. Serious comorbidities (chronic renal failure, hepatic disease, etc.) ;
3. Patients were on inhaled or oral mucolytics, or were receiving oxygen therapy or long-term oral antibiotics；
4. Poor compliance or cannot cooperate judged by doctors;
5. Participated in other clinical trials for nearly three months;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The age of all subjects are older than 18 . The diagnosis of bronchiectasis need reference to the guideline published by BTS in 2010 or 2012 China bronchiectasis expert consensus, clinical symptoms of cough and expectoration, with or without intermittent hemoptysis, and chest CT showed bronchiectasis there.All patients were clinically stable and had no evidence of exacerbation for at least 4 weeks before the study and had a negative history of allergy. None of patients had reversibility with inhaled salbutamol of 12% or more of predicted FEV1; All normal subjects had a negative history of allergy and normal lung function, they have no history of any lung disease (except for the history of pneumonia in the past time and small pulmonary nodules).
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Exhaled breath condensate pH and the disease severity | One year
  The Relationship between pH of exhaled breath condensate and disease severity of Bronchiectasis

SECONDARY OUTCOMES:
BSI scores | 30 days
  Assessment of the non-cystic fibrosis bronchiectasis severity according by the BSI score at the time of admission
SGRQ scores | 30 days
  Assessment of the quality of life of non-cystic fibrosis bronchiectasis according by the St.George respiratory questionnaire at the time of admission
Lung function (FEV1 %, FVC %, FEV1/FVC %) | One year
  Lung function will be measured at the time of admission
Sputum and peripheral blood inflammatory index (including IL-6, IL-8, IL-1β, TNF-a) | One year
  Sputum and peripheral blood inflammatory index will be assessed at the time of admission
Sputum neutrophil cell | One year
  Sputum neutrophil cell count and percentage will be assessed at the time of admission
Sputum bacteriological evaluation | One year
  Sputum bacteriological (pseudomonas aeruginosa and others) will be evaluated at the time of admission
Blood gases parameters （PaO2, SaO2, PaCO2, pH） | 30 days
  Blood gases will be assessed at the time of admission
Chest high-resolution computed tomography (CT) | One year
  Chest high-resolution computed tomography (CT) will be evaluated at the time of admission
Frequency of acute exacerbation during one year | 30 days
  The number of acute exacerbation will be recorded by telephone follow-up monthly. The definition of acute exacerbation: if there are at least one symptoms (increased sputum volume or purulent sputum, increased dyspnea, increased cough, lung function decline, increased fatigue) or new symptoms (fever, pleurisy, hemoptysis, require antimicrobial therapy), then prompted acute exacerbation.
Time to first exacerbation during the one-year follow up | 30 days
  The time to first exacerbation within one year after start of the study
The number of hospitalizations for exacerbation | 30 days
  The number of hospitalizations for exacerbation within one year after start of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jin-fu Xu, MD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital , Tongji University, Shanghai, Shanghai Municipality, China